CLINICAL TRIAL: NCT04586634
Title: Randomized Clinical Trial Assessing the Effect of Transanal Irrigation With Cone Catheter Versus Conservative Bowel Management on Symptoms of Low Anterior Resection Syndrome After Rectal Resection
Brief Title: Randomized Clinical Trial on Transanal Irrigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CP327
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2023-05

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peristeen (Active Comparator): Subjects to use newly developed Peristeen cone catherter device
  Interventions: Device: Peristeen cone catheter
- Standard of care (No Intervention): subjects continue with their standard of care treatment

INTERVENTIONS:
Device: Peristeen cone catheter — The active intervention is the Peristeen cone catheter device. The comparator in this investigation is current standard of care for patients with LARS which is conservative bowel management.
  Arms: Peristeen

SUMMARY:
Objective The primary objective is to demonstrate superiority of the Peristeen cone catheter compared to standard of care.

The secondary objective is to investigate quality of life and different benefits and aspects of treatment and satisfaction with the Peristeen cone catheter.

Design of the investigation This is a randomised, open-label, parallel investigation comparing the Peristeen cone catheter with standard of care in subjects with major LARS (LARS score ≥ 30). Each subject will be enrolled for a study duration of 12 weeks. Subjects will be randomized to the treatments stratified by neo-adjuvant radiotherapy.

The comparator in this study will be current standard of care for patients with LARS which is conservative bowel management. This is defined as: Supportive therapy according to the individual treatment protocols available at each participating site.

Primary endpoint and secondary endpoints

Primary endpoint:

• LARS score, obtained from the LARS score questionnaire*

Secondary endpoints:

* Number of subjects with Major LARS*
* FIQL Score - scale 1, Modified American Society for Colorectal Surgeons Questionnaire*
* FIQL Score - scale 2, Modified American Society for Colorectal Surgeons Questionnaire*
* FIQL Score - scale 3, Modified American Society for Colorectal Surgeons Questionnaire*
* FIQL Score - scale 4, Modified American Society for Colorectal Surgeons Questionnaire*
* EQ-5D-5L - utility score*
* EQ-5D-5L - VAS score (scale 0-10 cm)*
* Satisfaction with treatment (scale 0-10 cm)*
* Number of adverse events* *All endpoints are measured per subject at study completion

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age and have full legal Capacity
2. Have given written informed consent
3. Be mental and physical capable to perform transanal irrigation with cone catheter
4. Have a LARS score ≥ 30 after rectal resection
5. Be treated according to individual treatment protocol for conservatory bowel management at participating site
6. Have proof of complete healing of the anastomosis by endoscopy or radiology before stoma closure
7. At least 3-months from last surgery in colorectum
8. Be evaluated to be suitable for transanal Irrigation procedure with a cone catheter by endoscopy, defecography or comparable procedure

Exclusion Criteria:

1. Active/recurrent colorectal cancer
2. Leaking anastomosis
3. Known anal or colorectal stenosis
4. Within 4 weeks of endoscopic polypectomy
5. Ischaemic colitis
6. Acute inflammatory bowel disease
7. Acute diverticulitis
8. Current or planned pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Meurette, MD, Principal Investigator — CHU Nantes, France
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peristeen: Subjects to use newly developed Peristeen cone catherter device
  Peristeen cone catheter: The active intervention is the Peristeen cone catheter device.
  The comparator in this investigation is current standard of care for patients with LARS which is conservative bowel management.
Period: Overall Study
Arm/Group | Peristeen | Standard of Care
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Completed participants
Groups:
- Standard of Care: Subjects continue with their standard of care treatment which is conservative bowel management.
- Total: Total of all reporting groups
Arm/Group | Peristeen | Standard of Care | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (12.9) | 62.9 (10.1) | 63.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 13 | 9 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: LARS Score
Description: Obtained from the LARS score questionnaire on a scale from 0-42 in total score. Subscores are summed to get the total score. With 0 indicating lowest score and 42 highest score. 0-20 indicate No LARS, 21-29 minor LARS, 30-42 Major LARS.
Time Frame: Total score measured per subject at study completion after 12 weeks
Population: Missing data from 1 standard of care patient
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 14
score on a scale | 21.3 [14.7 to 27.8] | 32.2 [27.3 to 37.1]

2. Secondary Outcome: Number of Subjects With Major LARS
Description: as for outcome 1
Time Frame: 12 weeks
Population: missing data from 1 participant in standard of care
Measure: Count of Participants; unit: Participants
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 14
Participants | 5 | 10

3. Secondary Outcome: FIQL Score - Scale 1 Lifestyle, Modified American Society for Colorectal Surgeons Questionnaire
Description: The FIQL scale was thus interpreted for four scales exploring different aspects of the patient's quality-of-life. the Fecal Incontinence Quality of Life Scale (FIQL) contains 29 questions, across 4 domains, lifestyle (10 questions), Coping/Behavior (9 questions), Depression/Self Perception (7 questions), Embarrassment (3 questions).
  Items were scored 1 (least satisfactory quality-of-life) to 4 (most satisfactory quality-of-life) Results are reported as a Scale score which is the average (mean) response to all items in the scale (e.g., add the responses to all questions in a scale together and then divide by the number of items in the scale).
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 3.10 [2.65 to 3.55] | 2.60 [2.06 to 3.15]

4. Secondary Outcome: FIQL Score - Scale 2 Coping/Behavior, Modified American Society for Colorectal Surgeons Questionnaire
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 2.95 [2.55 to 3.35] | 2.37 [1.91 to 2.82]

5. Secondary Outcome: FIQL Score - Scale 3 Depression/Self-perception, Modified American Society for Colorectal Surgeons Questionnaire
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 3.41 [2.87 to 3.95] | 3.23 [2.76 to 3.71]

6. Secondary Outcome: FIQL Score - Scale 4 Embarrassment , Modified American Society For Colorectal Surgeons Questionnaire
Description: as for outcome 3
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 2.98 [2.57 to 3.38] | 2.76 [2.26 to 3.27]

7. Secondary Outcome: EQ-5D-5L - Utility Score
Description: Each of the five dimensions comprising the EQ-5D descriptive system (mobility, self-care, usual activates, pain/discomfort, anxiety/depression) was divided into five levels:
  1. no problem
  2. slight problems
  3. moderate problems
  4. severe problems
  5. unable to/extreme problems A unique health state was defined by combining one level from each of the five dimensions. i.e. state 12345 each state referred to by a 5-digit code was mapped into a utility score.
  Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead. EQ-5D-5L health states are converted into a single index 'utility' score using a scoring algorithm based on public preferences. Potential values from this algorithm can range from minus scores up to 1, in this case -0.525 to 1.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 0.92 [0.86 to 0.97] | 0.88 [0.81 to 0.95]

8. Secondary Outcome: EQ-5D-5L - VAS Score
Description: The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The VAS scale is from 0 to 100 with 0 indicating worst health and 100 best health possible.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 82.8 [70.2 to 95.5] | 71.4 [57.8 to 85.0]

9. Secondary Outcome: Satisfaction With Treatment
Description: Satisfaction with current bowel management treatment on a scale from 0 (total dissatisfaction) to 10 (perfect satisfaction)" rated on a VAS scale from 0 to 10 cm.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peristeen | Standard of Care
Number analyzed (Participants) | 15 | 15
score on a scale | 8.6 [7.4 to 9.7] | 5.9 [5.1 to 8.3]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Investigator Assessed at visits and phone calls
Arm/Group | Peristeen | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 5/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peristeen (N=16) | Standard of Care (N=16)
Mild Abdominal Pain (Gastrointestinal disorders) | 5 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT04586634/Prot_SAP_000.pdf